CLINICAL TRIAL: NCT06340594
Title: Single-stage Endoscopic Retrograde Cholangiopancreatography and Laparoscopic Cholecystectomy for Cholecystocholedocholithiasis: Which to Start With?
Brief Title: Single-stage ERCP and Laparoscopic Cholecystectomy for Cholecystocholedocholithiasis: Which to Start With?
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad Raafat, Lecturer at General surgery department, Assiut University
Other Study IDs: RF-2-2024
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Choledocholithiasis With Cholecystitis; Biliary Stones
Keywords: Choledocholithiasis; ERCP; Laparoscopic cholecystectomy; Cholecystocholedocholithiasis
MeSH Terms: conditions — Cholecystolithiasis; Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (ERCP 1st approach): The patients first underwent ERCP followed by standard 4 port LC.
  Interventions: Procedure: Laproscopic cholecystectomy (LC); Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP)
- Group B (LC 1st approach): The patients first underwent LC followed by ERCP.
  Interventions: Procedure: Laproscopic cholecystectomy (LC); Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Laproscopic cholecystectomy (LC) — Removal of gallbladder via laparoscopy
Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP) — Removal of bile duct stones via endoscopy

SUMMARY:
Chronic calculous cholecystitis is associated with common bile duct (CBD) stones in approximately 12% of patients. These patients need both cholecystectomy and CBD clearance of stones. The standard for cholecystectomy is laparoscopic cholecystectomy (LC) and the mostly common treatment used for CBD clearance is Endoscopic Retrograde Cholangiopancreatography (ERCP). The two interventions can be combined to be done at the same time under single anesthesia session. Studies of single stage ERCP+LC showed confirmed the safety and efficacy of the combined technique. However, some surgeons start with the ERCP while others start with LC.The aim of this study is to compare the start with ERCP followed by LC to the start with LC followed by ERCP when the two techniques are combined at the same session for treatment of chronic calculous cholecystitis associated with CBD stones regarding efficacy and safety of the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent single stage ERCP+LC for cholecystocholedocholithiasis

Exclusion Criteria:

* Contraindications to ERCP, or laparoscopic surgery
* Cholangitis and pancreatitis
* Previously failed ERCP

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic calculous cholecystitis associated with common bile duct (CBD) stones admitted in a tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Operative time operative time | time in minutes from intubation of the patient to the end of procedure
  total operative time of both ERCP+LC

SECONDARY OUTCOMES:
CBD clearance rate | up to 2 years
  success rate of retrieval of stones
Length of hospital stay | up to 2 weeks post-operative
  days of hospital stay
Mortality rate | up to 1 month postoperative
  number of deaths intraoperative and postoperative related to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine-Assiut University -Assiut-Egypt, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers SJ, Cello JP, Horn JK, Siperstein AE, Schecter WP, Campbell AR, Mackersie RC, Rodas A, Kreuwel HT, Harris HW. Prospective randomized trial of LC+LCBDE vs ERCP/S+LC for common bile duct stone disease. Arch Surg. 2010 Jan;145(1):28-33. doi: 10.1001/archsurg.2009.226. PMID 20083751
- [Background] Muhammedoglu B, Kale IT. Comparison of the safety and efficacy of single-stage endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy versus two-stage ERCP followed by laparoscopic cholecystectomy six-to-eight weeks later: A randomized controlled trial. Int J Surg. 2020 Apr;76:37-44. doi: 10.1016/j.ijsu.2020.02.021. Epub 2020 Feb 24. PMID 32105889
- [Background] Elgeidie A, Atif E, Elebidy G. Intraoperative ERCP for management of cholecystocholedocholithiasis. Surg Endosc. 2017 Feb;31(2):809-816. doi: 10.1007/s00464-016-5036-1. Epub 2016 Jun 22. PMID 27334962
- [Background] Williams EJ, Green J, Beckingham I, Parks R, Martin D, Lombard M; British Society of Gastroenterology. Guidelines on the management of common bile duct stones (CBDS). Gut. 2008 Jul;57(7):1004-21. doi: 10.1136/gut.2007.121657. Epub 2008 Mar 5. PMID 18321943
- [Background] Nie S, Fu S, Fang K. Comparison of one-stage treatment versus two-stage treatment for the management of patients with common bile duct stones: A meta-analysis. Front Surg. 2023 Feb 3;10:1124955. doi: 10.3389/fsurg.2023.1124955. eCollection 2023. PMID 36816010